CLINICAL TRIAL: NCT03816267
Title: Effectiveness of Salbutamol Administration by Nebulizer Versus Metered Dose Inhaler With Spacer in Acute Asthma in Children in Suez Canal University Hospital Emergency Department: A Randomized Control Trial
Brief Title: Salbutamol Administration by Nebulizer Versus Metered Dose Inhaler With Spacer in Asthma in Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Mona Azzam, Lecturer of Pediatrics, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3244
Record Dates: First submitted 2019-01-22; First posted 2019-01-25 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Bronchial Asthma
MeSH Terms: conditions — Asthma | interventions — Nebulizers and Vaporizers; Albuterol; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nebulizer (Active Comparator): Containing salbutamol
  Interventions: Device: Nebulizer; Drug: Salbutamol
- Metered Dose Inhaler and spacer (Experimental): Containing Salbutamol
  Interventions: Drug: Salbutamol; Device: Metered dose inhaler and spacer

INTERVENTIONS:
Device: Nebulizer — Nebulization via mask
  Arms: Nebulizer
Drug: Salbutamol — Delivery of appropriate dose according to weight
  Other Names: Albuterol, Ventolin
Device: Metered dose inhaler and spacer — Medication will be delivered through inhaler and spacer
  Other Names: MDI
  Arms: Metered Dose Inhaler and spacer

SUMMARY:
Asthma is a problem that affects many children and affects their physical health in addition to having a social and financial burden on individuals, families and healthcare systems. In our pediatric emergency department, nebulizers are still used for the management of asthma and, with the poor resources of families, they have no option of treatment at home. In this study, the investigators will compare the effectiveness of treatment through nebulizer versus metered dose inhaler and spacer in children with an acute asthmatic attack seeking medical care at the Pediatric Emergency Department of Suez Canal University Hospital.

DETAILED DESCRIPTION:
Primary Objective:

To determine whether the administration of a B2 agonist by metered dose inhaler with spacer is as effective as the administration of B2 agonist by nebulizer for the treatment of an acute asthmatic episode in children seeking medical care in the Pediatric Emergency Department of Suez Canal University Hospital.

Secondary Objectives:

1. Comparison of patients' visit duration in the ER room between the two groups.
2. Comparison of hospitalization rate between the two groups.
3. Comparison of parent/patient satisfaction between the two groups. Study design Single-blinded randomized control trial.

Study location This study will be conducted in the Pediatric Emergency Department in Suez Canal University Hospital.

Study population This study will include patients presenting with an acute exacerbation of asthma at the Pediatric Emergency Department in Suez Canal University Hospital starting July 2017 until our sample size is fulfilled.

Inclusion criteria:

Children ranging from 2 - 14 years old. Both genders will be included. Patients with an acute exacerbation of asthma.

Exclusion criteria:

Patients with arrhythmia and cardiac diseases. Patients with thyroid diseases. Patients with bronchiolitis, pneumonia. Patients with status asthmaticus requiring immediate pediatric intensive care unit hospitalization.

Sampling All children fulfilling the inclusion criteria will be included consecutively until the calculated sample size has been reached.

Sample size

The sample size will be calculated using the following formula:

(Dawson & Trapp, 2004)

Where:

n= sample size Zα/2 = 1.96 (The critical value that divides the central 95% of the Z distribution from the 5% in the tail) Zβ = 0.84 (The critical value that separates the lower 20% of the Z distribution from the upper 80%) σ = the estimate of the standard deviation = 1.5 (Rubilar et al., 2000) µ1 = mean in the nebulizer group = 4.4 (Rubilar et al., 2000) µ2 = mean in the metered-dose inhaler group = 3.3 (Rubilar et al., 2000) So, by calculation, the sample size will be equal to 30 cases per group, giving a total sample size of 60 cases.

Methods of data collection

Infants and children known to have asthma coming to the Pediatric Emergency Department of Suez Canal University Hospital and fulfilling the inclusion criteria will be assessed according to the following clinical respiratory score:

(Mild 0-3 moderate 4-7 severe 8-12)17

The target population is patients who presented with moderate to severe wheezing (score 4-12).

Randomization will take place through an online program for randomization of clinical trials. The patients will be divided into two groups, one of them treated by the available nebulizer and the other by MDI with spacer. The investigators cannot blind patients to the treatment as there is an obvious difference between the two modalities.

However, the assessment of the respiratory score before and after the treatment will be performed by an independent physician who will not be involved in the decision-making and randomization of treatment. This physician will be asked to assess initially and then reassess after the equipment has been removed to avoid any bias.

Dosage and administration:

The nebulizer group will receive salbutamol aerosol solution (0.25 mg/kg weight, up to a maximum of 5 mg in 3.5 mL of normal saline solution. Aerosols will be generated by jet nebulizers powered by oxygen and delivered via a face mask for 7 min every 20 min during the first hour (a total of three nebulizations/hr.). A flow rate of 7 L/min will be used.

The metered dose inhaler with spacer group will receive two puffs of salbutamol (100 mcg/puff) every 10 min 5 times over 1 hr. (a total of 10 puffs/hr.), using a spacer device with a face mask. Following each puff, the children will take breaths for a full minute from the spacer device held in place.

Assessment:

Patients will be reassessed after one hour and score <4 is considered a success while score>4 is failure of therapy.

Patients of same degree of severity of the attack will be compared together according to the following characteristics: duration of treatment preparation and delivery, clinical outcome, patient satisfaction after use and hospitalization rate.

Each patient will have a form: Page 1 will be an informed consent to be signed before randomization of treatment. Page 2 will include the following items

1. personal data (name, age, address, telephone number to be in contact with the patient and know if there were repeated visits after this attack within the same week). In addition, the researcher's phone number will be accessible to the patients.
2. Medical history (other illnesses, medications, degree of asthma either intermittent or persistent)
3. Clinical assessment (clinical respiratory score before and after treatment)
4. Patient satisfaction with given modality on a Likert scale from 1-5. This will be asked by the blinded assessor and will include questions regarding:

   * Comfort with modality used
   * Duration of modality used
   * Ease of administration
   * Confidence in repeating treatment on their own at home if required

ELIGIBILITY:
Inclusion Criteria:

* Children ranging from 2 - 14 years old.
* Both genders will be included.
* Patients with an acute exacerbation of asthma.

Exclusion Criteria:

* Patients with arrhythmia and cardiac diseases.
* Patients with thyroid diseases.
* Patients with bronchiolitis, pneumonia. Patients with status asthmaticus requiring immediate pediatric intensive care unit hospitalization.

Ages: 2 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-03-15 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical improvement | 1 hour
  Clinical respiratory score change (see Study Protocol for details)

SECONDARY OUTCOMES:
Rate of Hospitalization | 4 hours
  Admission into inpatient or intensive care unit
Patient satisfaction | 1 hour
  Patient or parent satisfaction using Likert scale (see Study Protocol for details)

CONTACTS AND LOCATIONS:
Overall Officials: Alaa Zeitoun, Prof, Study Chair — Suez Canal University
Locations (1):
- Suez Canal University Hospital, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rubilar L, Castro-Rodriguez JA, Girardi G. Randomized trial of salbutamol via metered-dose inhaler with spacer versus nebulizer for acute wheezing in children less than 2 years of age. Pediatr Pulmonol. 2000 Apr;29(4):264-9. doi: 10.1002/(sici)1099-0496(200004)29:43.0.co;2-s. PMID 10738013

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT03816267/Prot_SAP_000.pdf